CLINICAL TRIAL: NCT04957290
Title: A Phase 1b/2a Multicenter Study of NOX66 and External Beam Radiotherapy in Patients With Metastatic Castration-resistant Prostate Cancer and Other Solid Tumors
Brief Title: A Study of NOX66 and External Beam Radiotherapy in Patients With Metastatic Castration-resistant Prostate Cancer and Other Solid Tumors
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Slow Recruitment
Sponsor: Noxopharm Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NOX66-005
Record Dates: First submitted 2021-06-16; First posted 2021-07-12 (Actual); Results first posted 2024-06-18 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-05

CONDITIONS: Metastatic Castration-resistant Prostate Cancer and Other Solid Tumors
Keywords: Dose Escalation; Dose Expansion; Prostate-specific antigen; Maximum tolerated dose; Recommended Phase 2 dose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Part 1: Dose Cohort 1: NOX66 800 mg (Experimental)
  Interventions: Drug: NOX66; Radiation: EBRT
- Part 1: Dose Cohort 2: NOX66 1200 mg (Experimental)
  Interventions: Drug: NOX66; Radiation: EBRT
- Part 1: Dose Cohort 3: NOX66 1600 mg (Experimental)
  Interventions: Drug: NOX66; Radiation: EBRT
- Part 1: Dose Cohort 4: NOX66 2400 mg (Experimental)
  Interventions: Drug: NOX66; Radiation: EBRT
- Part 2: Arm 1: Patients with mCRPC (RP2D NOX66) (Experimental)
  Interventions: Drug: NOX66; Radiation: EBRT
- Part 2: Arm 2: Patients with BC or NSCLC (RP2D NOX66) (Experimental)
  Interventions: Drug: NOX66; Radiation: EBRT

INTERVENTIONS:
Drug: NOX66 — NOX66 800 mg daily (400 mg suppository twice daily [BID]).
  Arms: Part 1: Dose Cohort 1: NOX66 800 mg
Drug: NOX66 — NOX66 1200 mg daily (600 mg suppository BID).
  Arms: Part 1: Dose Cohort 2: NOX66 1200 mg
Drug: NOX66 — NOX66 1600 mg daily (800 mg suppository BID).
  Arms: Part 1: Dose Cohort 3: NOX66 1600 mg
Drug: NOX66 — NOX66 2400 mg daily (1200 mg suppository BID).
  Arms: Part 1: Dose Cohort 4: NOX66 2400 mg
Drug: NOX66 — NOX66 RP2D
  Arms: Part 2: Arm 1: Patients with mCRPC (RP2D NOX66); Part 2: Arm 2: Patients with BC or NSCLC (RP2D NOX66)
Radiation: EBRT — The dose levels of EBRT will be either 8 Gy as a single fraction, or 20/25 Gy as 5 fractions given over 5 to 10 days.

SUMMARY:
This is a Phase 1b/Phase 2a, open-label, multicenter study to determine the safety, tolerability, recommended Phase 2 dose (RP2D), efficacy, pharmacokinetics (PK) and pharmacodynamic (PD) properties of idronoxil when rectally administered as a suppository (NOX66) to patients with any solid tumor (Part 1) and patients with metastatic castration-resistant prostate cancer (mCRPC), breast cancer (BC) and non-small-cell lung cancer (NSCLC) (Part 2) who are eligible for low-dose external beam radiotherapy (EBRT) for at least one symptomatic or minimally symptomatic lesion (for the prevention of symptoms).

DETAILED DESCRIPTION:
The study is divided into 2 parts: Part 1 (dose escalation) and Part 2 (dose expansion). The study design allows an exploration of different doses of NOX66 (800 mg, 1200 mg, 1600 mg and 2400 mg) with safety monitoring to ensure the safety of the patients. In Cycle 1, NOX66 will be administered for 14 days followed by a 7-day rest period on a 21-day cycle. From Cycle 2 onwards, NOX66 will be administered for 7 days followed by a 7-day rest period on a 14-day cycle. Patients will continue to receive NOX66 on a cyclical basis until disease progression, unacceptable toxicity, withdrawal of consent, start of a new anticancer therapy, withdrawal of the patient by the Investigator or the end of study is reached.

ELIGIBILITY:
Inclusion Criteria:

* Patient has a minimum life expectancy of 6 months
* Histological or cytological confirmation of prostate cancer, BC, NSCLC and any other solid tumors
* Confirmed metastatic disease by imaging
* Documented disease progression following first or later lines of anticancer systemic treatment
* Patient is eligible for low-dose EBRT for at least one lesion
* Patients with prior RT are eligible, only if there is no potential for field overlap between the prior RT and the planned RT
* For patients with BC or NSCLC: Patient must have at least one measurable lesion as per RECIST v1.1 (in Part 2 only)
* Patient has ECOG performance status of 0 to 2
* Adequate bone marrow, renal, and liver function
* Metastatic Castration-resistant Prostate Cancer: Baseline testosterone levels ≤ 14.4 ng/dL and ongoing medical castration must be maintained throughout the duration of the study; patient has evidence of symptomatic and/or progressive disease
* Breast Cancer Patients: Known hormone receptor status (estrogen receptors/progesterone receptors or estrogen receptors alone). Breast cancer patients are allowed to be on background hormonal treatment.

Exclusion Criteria:

* Patient has tumor involvement of the central nervous system
* Impaired cardiac functioning or clinically significant cardiac disease
* Uncontrolled hypertension despite two concomitant antihypertensive therapies
* Patients who have had a colectomy (total or left hemicolectomy) with re-anastomosis
* Patients for whom administration of the suppositories are likely to cause pain or difficulties in absorption
* Patients with fecal impaction or uncontrolled irritable bowel disease
* Patients with inflammatory bowel disease
* Any other disease, metabolic dysfunction, physical examination finding or clinical laboratory finding that, in the Investigator's opinion, gives reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug, may affect the interpretation of the results, render the patient at high risk from treatment complications or interferes with obtaining informed consent
* Patients with oligometastatic disease (fewer than 5 metastatic lesions) amenable to standard therapy will be excluded
* Patients who have had RT to the region of the rectum or will require RT to the region of the rectum during the trial
* Uncontrolled active infection requiring intravenous antibiotic, antiviral or anti-fungal medications within 14 days before the first dose administration
* Receiving or having received anticancer treatment
* Patient has received corticosteroids at a dose of > 10 mg prednisone/day or equivalent for any reason within 4 weeks prior to receiving the first dose administration
* Patient is not willing to use suppositories
* Patient has a positive reverse transcription polymerase chain reaction (RT-PCR) test for severe acute respiratory coronavirus 2 (SARS-CoV-2) prior to Screening or enrollment, or has clinical signs and symptoms consistent with SARS-CoV-2 infection; e.g., fever, dry cough, dyspnea, sore throat, fatigue or positive SARS-CoV-2 test result within 2 weeks prior to Screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2021-10-25 (Actual); Primary Completion 2023-05-10 (Actual); Study Completion 2023-06-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Beverly Hills Cancer Center, Beverly Hills, California
  - The University of Texas - MD Anderson Cancer Center - Genitourinary (GU) Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 21 patients
Period: Overall Study
Arm/Group | Part 1: Dose Cohort 1: NOX66 800 mg | Part 1: Dose Cohort 2: NOX66 1200 mg | Part 1: Dose Cohort 3: NOX66 1600 mg | Part 1: Dose Cohort 4: NOX66 2400 mg | Part 2: Arm 1: Patients With mCRPC (RP2D NOX66) | Part 2: Arm 2: Patients With BC or NSCLC (RP2D NOX66)
Started | 4 | 7 | 10 | 0 (cohort 4 never started) | 0 (Part 2 never started) | 0 (Part 2 never started)
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 4 | 7 | 10 | 0 | 0 | 0
Not completed — Progressive disease | 3 | 3 | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 0 | 0 | 0
Not completed — Death | 0 | 2 | 1 | 0 | 0 | 0
Not completed — non compliance with study drug | 0 | 1 | 0 | 0 | 0 | 0
Not completed — none specified. | 0 | 1 | 2 | 0 | 0 | 0
Not completed — unacceptable toxicity | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 0
Not completed — study terminated by sponsor | 0 | 0 | 2 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Study terminated early during part 1- cohort 3.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: Dose Cohort 1: NOX66 800 mg | Part 1: Dose Cohort 2: NOX66 1200 mg | Part 1: Dose Cohort 3: NOX66 1600 mg | Part 1: Dose Cohort 4: NOX66 2400 mg | Part 2: Arm 1: Patients With mCRPC (RP2D NOX66) | Part 2: Arm 2: Patients With BC or NSCLC (RP2D NOX66) | Total
Number analyzed (Participants) | 4 | 7 | 10 | 0 | 0 | 0 | 21
Age, Continuous [Median (Full Range); unit: years] | 69 [60 to 80] | 73 [51 to 82] | 67.5 [27 to 93] |  |  |  | 68 [27 to 93]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 1 |  |  |  | 5
  Male | 1 | 6 | 9 |  |  |  | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 3 |  |  |  | 7
  Not Hispanic or Latino | 2 | 5 | 7 |  |  |  | 14
  Unknown or Not Reported | 0 | 0 | 0 |  |  |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 |  |  |  | 1
  Asian | 0 | 0 | 0 |  |  |  | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 |  |  |  | 0
  Black or African American | 1 | 2 | 0 |  |  |  | 3
  White | 3 | 5 | 9 |  |  |  | 17
  More than one race | 0 | 0 | 0 |  |  |  | 0
  Unknown or Not Reported | 0 | 0 | 0 |  |  |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 6 | 8 |  |  |  | 18
  Australia | 0 | 1 | 0 |  |  |  | 1
  Hungary | 0 | 0 | 2 |  |  |  | 2

OUTCOME MEASURES:

1. Primary Outcome: Part 1 (Dose Escalation): Number of Dose-limiting Toxicities (DLTs)
Description: Maximum tolerated dose (MTD) and RP2D of NOX66 in combination with low-dose EBRT in patients with any solid tumor. MTD is defined as the dose level at which no more than 1 patient out of 6 has a DLT at the end of Cycle 1. RP2D is the highest dose at which no more than 1 patient out of 6 has a DLT at the end of Cycle 1 and the dosage form, is acceptable to patients.
  A DLT is defined as an AE that occurs during Cycle 1 (Day 1 to Day 21) that is unrelated to the disease, intercurrent illness or concomitant medications and that, possibly- definitely related to NOX66 alone or in combination with EBRT:
  Grade (G) ≥3 non-hematological toxicity; G≥3 febrile neutropenia; G4 thrombocytopenia > 5 days; G3 thrombocytopenia with bleeding or in combination with a G ≥3 blood and lymphatic system disorder.; G3 AST or ALT that is + a ≥G2 rise in bilirubin >7 days; AST or ALT > 8 × ULN; AE causing treatment delay > 14 days.
Time Frame: Cycle 1 (Day 1 to Day 21)
Population: All patients that completed cycle 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Dose Cohort 1: NOX66 800 mg | Part 1: Dose Cohort 2: NOX66 1200 mg | Part 1: Dose Cohort 3: NOX66 1600 mg
Number analyzed (Participants) | 4 | 7 | 10
Participants | 0 | 0 | 0

2. Secondary Outcome: Part 1: Incidence of Adverse Events (AEs) for NOX66
Description: Characterization of the safety and tolerability of NOX66.
Time Frame: From Screening (Days -28 to -2) until the Follow-up visit/End of Study (EOS) (through study completion, an average of 19 month)
Population: Safety population = all participants who received at least one dose of NOX66
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Dose Cohort 1: NOX66 800 mg | Part 1: Dose Cohort 2: NOX66 1200 mg | Part 1: Dose Cohort 3: NOX66 1600 mg
Number analyzed (Participants) | 4 | 7 | 10
Participants
  With at least one Adverse Event | 4 | 7 | 9
  With at least one TEAE (Treatment Emergent Adverse Event) | 4 | 7 | 9
  Dose Limiting Toxicity | 0 | 0 | 0
  Fatal TEAE | 0 | 1 | 0
  AEs that were greater than Grade 2 severity | 1 | 5 | 5
  TEAE related to Study Treatment (NOX66) | 4 | 4 | 6

3. Secondary Outcome: Part 1: TEAEs by Relationship to EBRT Administration
Description: Evaluation of the safety and tolerability of both doses of EBRT (8 Gy or 20/25 Gy).
Time Frame: From Screening (Days -28 to -2) until the Follow-up visit/EOS (through study completion, an average of 19 month)
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Dose Cohort 1: NOX66 800 mg | Part 1: Dose Cohort 2: NOX66 1200 mg | Part 1: Dose Cohort 3: NOX66 1600 mg
Number analyzed (Participants) | 4 | 7 | 10
Participants
  Possibly Related | 1 | 2 | 3
  Related | 0 | 2 | 2
  No AEs related to EBRT | 3 | 3 | 5

ADVERSE EVENTS:
Time Frame: All AEs and SAEs will be collected from the signing of the ICF until 30 days after the last dose of study drug at the time points specified in the Schedule of assessments with an average of 7 months for each participant.
Arm/Group | Part 1: Dose Cohort 1: NOX66 800 mg | Part 1: Dose Cohort 2: NOX66 1200 mg | Part 1: Dose Cohort 3: NOX66 1600 mg
All-Cause Mortality (participants affected / at risk) | 0/4 | 2/7 | 1/10
Serious Adverse Events (participants affected / at risk) | 1/4 | 3/7 | 5/10
Other Adverse Events (participants affected / at risk) | 4/4 | 6/7 | 9/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Dose Cohort 1: NOX66 800 mg (N=4) | Part 1: Dose Cohort 2: NOX66 1200 mg (N=7) | Part 1: Dose Cohort 3: NOX66 1600 mg (N=10)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Dose Cohort 1: NOX66 800 mg (N=4) | Part 1: Dose Cohort 2: NOX66 1200 mg (N=7) | Part 1: Dose Cohort 3: NOX66 1600 mg (N=10)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 4 (5)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)
Anorectal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Proctitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 3 (4)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 2 (3)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (4)
Fatigue (General disorders) | 1 (1) | 2 (2) | 2 (3)
Lymphopenia (Blood and lymphatic system disorders) | 2 (2) | 1 (6) | 1 (2)
Anaemia (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 1 (4)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (4)

LIMITATIONS AND CAVEATS:
Dose escalation progressed through the first 3 planned dose levels before the Sponsor decided to terminate the study for business reasons; the decision was not based on any safety concerns with NOX66.

Due to early termination, none of the efficacy parameters were able to be measured therefore only safety outcomes are available.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan: Latest approved version (2022-11-23): https://cdn.clinicaltrials.gov/large-docs/90/NCT04957290/Prot_SAP_000.pdf
  • Study Protocol and Statistical Analysis Plan: version for first patient enrolled (2022-01-21): https://cdn.clinicaltrials.gov/large-docs/90/NCT04957290/Prot_SAP_001.pdf